CLINICAL TRIAL: NCT05391399
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial Evaluating the Safety and Efficacy of Interlocking Detachable Coils System for Embolization of Peripheral Arterial
Brief Title: Use of Interlocking Detachable Coils System in Embolization of Peripheral Arterial Embolization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Shenqi Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP01-025A
Record Dates: First submitted 2022-05-22; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A Interlocking detachable coils system (Experimental): The coil is designed with mechanical release, which can be recovered and repositioned at any time when the release process meets certain conditions.
  Interventions: Device: Interlocking detachable coils system
- group B Interlock Fibered IDC Occlusion System (Active Comparator): The coil adopts the design of mechanical release, and can be recovered, repositioned and released at any time when the release process meets certain conditions.
  Interventions: Device: Interlock Fibered IDC Occlusion System

INTERVENTIONS:
Device: Interlocking detachable coils system — Mainly used to block or slow blood flow in the peripheral vascular system during embolization procedures.
  Arms: group A Interlocking detachable coils system
Device: Interlock Fibered IDC Occlusion System — Mainly used to block or slow blood flow in the peripheral vascular system during embolization procedures.
  Arms: group B Interlock Fibered IDC Occlusion System

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of interlocking detachable coils system in the treatment of Chinese patients with embolization of peripheral arterial in comparison with Interlock Fibered IDC Occlusion System

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, non-inferiority, randomized controlled clinical trial. The plan is to recruit patients with peripheral arterial disease requiring embolization and then perform peripheral arterial embolization based on randomization using devices in the experimental group or control group. This trail will be conducted in a number of experimental institutions in China, and a total of 116 subjects are planned to be enrolled. All subjects were treated with the interlocking detachable coils system and were evaluated during surgery and before discharge from the treatment of experimental or control devices, followed up at 1 month, 3 months, and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years;
2. Subject diagnosed with peripheral arterial embolization by preoperative imaging (CTA);
3. The target vessel can be embolized in one operation;
4. The visual diameter of the target blood vessel is 5mm-30mm;
5. Subjects or their legal representatives can understand the purpose of the trial, voluntarily participate and sign the written informed consent, and can be followed up.

Exclusion Criteria:

1. Definite allergy, resistance or contraindication to antiplatelet agents, anticoagulants, contrast agents and/or anesthetics;
2. Definite allergy to platinum, tungsten and/or any substance in the test coil;
3. Subjects are not suitable for anesthesia or endovascular surgery, such as those with severe respiratory, heart, lung, liver, kidney disease or coagulation disorders (such as hemophilia);
4. The target vessel has undergone previous surgery and/or major cardiovascular surgery within 3 months;
5. The target aneurysm is dissecting aneurysm, infected aneurysm, ruptured aneurysm, and aneurysm caused by connective tissue disease;
6. Women who are pregnant or breastfeeding;
7. Subjects who are participating in clinical trials of other drugs or devices that have not reached the end point of the trial;
8. The researcher believes that it is not suitable to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
target vessel occlusion rate | 6 months
  no blood flow through the occluded segment of the target vessel

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No